CLINICAL TRIAL: NCT06890052
Title: Effects of Isolated Lumbar Extension Resistance Exercise and the Impact of Additional Treatments on Multifidus Muscle Morphology, Strength, and Patient-Reported Outcomes in Chronic Low Back Pain and Radiculopathy Related to Spinal Disorders: a Closely-Monitored Clinical Trial
Brief Title: Effects of Isolated Lumbar Extension Resistance Training Alone and in Combination with General Exercise and Manual Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Collaborators: Private Spine Center Dr. Alfen (Unknown)
Responsible Party: Principal Investigator, Bruno Domokos, Project Coordinator, University of Wuerzburg
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01/2023
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Multifidus; Exercise Therapy; Diagnostic Imaging
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ILEX-Only (Active Comparator): A supervised 16-week program consisting of 25 sessions of isolated lumbar extension resistance exercise (ILEX) using a new machine-based device. The program includes two sessions per week for the first nine weeks, followed by one session per week for the remaining seven weeks.
  Interventions: Other: Targeted exercise program
- ILEX supplemented with General Exercise and Manual Therapy (Experimental): A supervised 16-week program consisting of 25 sessions of isolated lumbar extension resistance exercise (ILEX) using a new machine-based device. The program includes two sessions per week for the first nine weeks, followed by one session per week for the remaining seven weeks. Each session is supplemented with four general strengthening exercises. Additionally, patients receive manual therapy (MT).
  Interventions: Other: Targeted exercise as part of an integrative therapy program

INTERVENTIONS:
Other: Targeted exercise program — Participants in the active comparator group will perform 25 sessions of isolated lumbar extension resistance exercise (ILEX) using a new machine-based device equipped with a pelvic restraint system to ensure targeted conditioning of the paraspinal muscles. The exercise will be supplemented by visual biofeedback displayed on a computer screen. A detailed protocol will be followed, incorporating an individualized, diagnosis-based range of motion and progressive resistance overload. The supervised 16-week program consists of two sessions per week for the first nine weeks, followed by one session per week for the remaining seven weeks.
  Arms: ILEX-Only
Other: Targeted exercise as part of an integrative therapy program — Participants in the experimental group will perform 25 sessions of isolated lumbar extension resistance exercise (ILEX) using a new machine-based device equipped with a pelvic restraint system to ensure targeted conditioning of the paraspinal muscles. The exercise will be supplemented by visual biofeedback displayed on a computer screen.
  A detailed protocol will be followed, incorporating an individualized, diagnosis-based range of motion and progressive resistance overload.
  The supervised 16-week program consists of two sessions per week for the first nine weeks, followed by one session per week for the remaining seven weeks.
  Each session is supplemented with general exercises for the back and trunk muscles (e.g., lat pulldown, abdominal crunch). In addition, participants will receive at least five sessions of therapy, which may include joint mobilization, tissue treatment, stress management, and other therapeutic modalities.
  Arms: ILEX supplemented with General Exercise and Manual Therapy

SUMMARY:
This study examines effects of machine-based isolated lumbar extension resistance exercise (ILEX) on paraspinal muscle morphology and function, as well as pain intensity, disability and quality of life in patients with chronic low back pain and radiculopathy related to specific spinal disorders. Current guidelines emphasize the necessity of treating chronic low back pain with integrative, holistic approaches due to its multidimensional nature. At the same time, an increasing number of studies highlight the importance of restoring lumbar muscle function and morphology through targeted training. Regarding ILEX, existing studies already support its clinical value, however, the optimal integration of ILEX with other therapeutic modalities remains unclear.

Two groups will be enrolled in an ILEX protocol (16 weeks, 25 sessions), while one of the groups will additionally participate in general exercise and manual therapy.

After completion of the main program, participants will be given different options to continue the exercise therapy with a reduced frequency (e.g., once per month). After six months, a follow-up assessment will be conducted with all participants to analyze long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. chronic LBP for > 3 months, defined as pain in the region between the lower ribs and gluteal folds, with or without leg pain
2. seeking care in the facility of the study
3. doctoral assessment indicating symptoms related to disc herniations/protrusions and other specific conditions
4. moderate pain levels at the time of doctoral assessment

Exclusion Criteria:

1. acute low back pain (pain < 3 months)
2. familiarity with the device (usage within the previous 12 months)
3. fractures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
Multifidus cross-sectional area (CSA; cm2) | Baseline, 3-week, 6-week, 9-week, 16-week
  Multifidus muscle cross-sectional area measurements are obtained from ultrasound (US) from the L4/L5 spinal level (left and right)
Multifidus muscle thickness (MT; cm) | Baseline, 3-week, 6-week, 9-week, 16-week
  Multifidus muscle thickness is measured with ultrasound (US) from the L4/L5 spinal level (left and right)
Multifidus echo intensity (EI; 0 -255 AU) | Baseline, 3-week, 6-week, 9-week, 16-week
  Multifidus echo intensity (EI) is measured with ultrasound (US) from the cross-sectional area of the L4/L5 spinal level (left and right). EI is measured in arbitrary units (AU) via ImageJ on a scale from 0 (black) to 255 (white)

SECONDARY OUTCOMES:
Pain intensity (0-100) | Baseline, 3-week, 6-week, 9-week, 16-week
  Pain intensity is measured with the visual analog scale (VAS) on a rating scale from 0 (no pain) to 100 (maximum pain).
Disability (0-50) | Baseline, 3-week, 6-week, 9-week, 16-week
  Disability in relation to LBP is measured with the Oswestry Disability Index (ODI). It includes 10 items (e.g., sitting, standing, personal care) with a range from 0-6 with higher scores indicating greater disability.
Health-related quality of life (QoL; 0-100) | Baseline, 3-week, 6-week, 9-week, 16-week
  Health-related quality of life (QoL) is measured with the short-form survey 345 (SF-36). The survey consists of 8 domains assessing physical and mental sum scores (PCS and MCS). Scores in each domain can range from 0 (zero health) to 100 (perfect health).
Isometric Lumbar Extensor Muscle Strength (Nm) | Baseline, 3-week, 6-week, 9-week, 16-week
  Isometric lumbar extensor strength is measured with an isokinetic dynamometer as part of the Powerspine Back ILEX device. Measurements were taken at 39°, 30°, 24° and 15° in Newton meter (Nm).
Postural Alignment (°) | Baseline, 3-week, 6-week, 9-week, 16-week
  Postural alignment will be measured with an infrared-based surface scanner (IDIAG M360). Included measures are angulations of 1) the thoracic spine, 2) the lumbar spine, and 3) the sacral inclination.
Mobility (°) | Baseline, 3-week, 6-week, 9-week, 16-week
  Mobility is measured with an infrared-based surface scanner (IDIAG M360). Included measures are the mobility of the thoracic spine, the lumbar spine and the sacral inclination.
Stability (°) | Baseline, 3-week, 6-week, 9-week, 16-week
  Stability is measured with an infrared-based surface scanner (IDIAG M360) and application of the Mathiass' Test. Included measures are angulations the thoracic spine, the lumbar spine, and the sacral inclination.
Muscle activity in sitting posture (mV) | Baseline, 3-week, 6-week, 9-week, 16-week
  Sitting posture activity at the L4/L5 lumbar segment (bilateral) is measured using surface electromyography.
Muscle activity during static contraction in prone position (mV) | Baseline, 3-week, 6-week, 9-week, 16-week
  Muscle activity during static contractin in prone position is measured at the L4/L5 level (bilateral) using surface electromyography.
Muscle activity during standing dynamic forward bend (mV) | Baseline, 3-week, 6-week, 9-week, 16-week
  Muscle activity during during standing dynamic forward bend is measured at the L4/L5 level (bilateral) using surface electromyography.
Heart rate variability (HR, RSA, RMSSD) | Baseline, 3-week, 6-week, 9-week, 16-week
  Measures of heart rate variability are obtained including heart rate (beats/minute), respiratory sinus arrhytmia (RSA) and root mean square of successive differences (RMSSD).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Raschka, Prof. Dr. Dr. Dr., Study Director — University of Wuerzburg
Locations (1):
- University of Wuerzburg, Institute of Sports Science, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Domokos B, Domokos J, Andersson G, Mannel S, Weigel LM, Koch HJ, Wallmann-Sperlich B, Raschka C, Spang C. Isolated lumbar extension exercise alone or in a multimodal program for low back pain and radiculopathy: a non-randomized controlled trial. Sci Rep. 2025 Oct 23;15(1):37157. doi: 10.1038/s41598-025-22452-x. PMID 41131158
- See also: Are the size and composition of the paraspinal muscles associated with low back pain? A systematic review — https://pubmed.ncbi.nlm.nih.gov/28756299/
- See also: Isolated Lumbar Extension Resistance Exercise in Limited Range of Motion for Patients with Lumbar Radiculopathy and Disk Herniation-Clinical Outcome and Influencing Factors — https://pubmed.ncbi.nlm.nih.gov/34070780/
- See also: A review of the specificity of exercises designed for conditioning the lumbar extensors — https://pubmed.ncbi.nlm.nih.gov/24092889/
- See also: The Effects of Combined Motor Control and Isolated Extensor Strengthening versus General Exercise on Paraspinal Muscle Morphology, Composition, and Function in Patients with Chronic Low Back Pain: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/37762861/